CLINICAL TRIAL: NCT05293457
Title: A Prospective Multicenter Study of AI-assisted Gastroscopic Varices Diagnosis
Brief Title: AI-assisted Gastroscopic Varicose Vein Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, ChenMingkai, Clinical Professor, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2022-K014
Record Dates: First submitted 2022-02-13; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Artificial Intelligence
Keywords: artificial intelligence; Varicose veins; Cirrhosis
MeSH Terms: conditions — Varicose Veins; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of the accuracy of AI in assisting gastroscopic varices diagnosis through a prospective multicenter study

DETAILED DESCRIPTION:
This study is a multi-center prospective study. Patients who meet the inclusion and exclusion criteria of the study will collect their basic information during outpatient and hospitalization. The designated doctor will introduce the significance of this study to the patients and sign the informed consent. After the endoscopy of the patient, the video of the operation under the endoscope was collected and saved, and the AI was imported to obtain its conclusions on the above characteristics, as well as stratification and treatment recommendations. Follow-up requirements for third-party physicians who meet the inclusion criteria, record their various diagnosis and treatment recommendations after watching the video (mainly in the form of a selection questionnaire to avoid subjective bias), and the content of the questionnaire includes the veins observed in the endoscopic operation video. Varicose related features (with or without red sign, bleeding sign, varicose vein shape, diameter, color, mucosal sign), and corresponding risk stratification and treatment recommendations are required. For videos with inconsistent conclusions between AI and physicians, physicians will be asked to watch these videos with AI prompts again to give their opinions, and there will be a two-week buffer period between the first time and the second viewing. The reference standard for diagnosis will be obtained by three endoscopists watching videos without AI prompts, and the conclusions drawn by the three experts will be used as the reference standard. When the three experts have inconsistent conclusions, the three experts will discuss A consensus shall prevail. If no consensus can be reached in the end, the video will be discarded.

Primary and secondary endpoints were obtained by comparing the accuracy of diagnosis made by physicians and AI. All data were analyzed by SPSS statistical software.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or above;
2. Gastroscopy and related examinations are required to further clarify the characteristics of digestive tract diseases;
3. Patients with liver cirrhosis who have signs or symptoms of portal hypertension and have clinical indications for endoscopic screening for varicose veins.
4. Able to read, understand and sign the informed consent;
5. The researcher believes that the subjects can understand the process of the clinical study, are willing and able to complete all the research procedures and follow-up visits, and cooperate with the research procedures.

Exclusion Criteria:

1) Pregnant or breastfeeding women; 2) Patients with a history of esophagogastric surgery; 3) Patients who have received interventional or endoscopic treatment in the past; 4) The patient has high-risk diseases or other special conditions that are not suitable for participating in clinical trials; 5) The patient is clearly diagnosed with esophageal or gastric diverticulum, polyps, cancer and other diseases that may affect the observation of varicose veins; 6) The patient's endoscopic video cannot reach a consensus diagnosis and treatment opinion after being watched by three experts.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis who visited each center of the study from February 2022 to December 2022.
Sampling Method: Probability Sample
Enrollment: 793 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2022-10-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
The accuracy of artificial intelligence | 2022/12/25
  Accuracy of AI in the description and treatment recommendations of esophagogastric varices diagnosis and endoscopic findings (form, color, red sign, hemorrhagic sign, and mucosal findings).

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT05293457/Prot_000.pdf